CLINICAL TRIAL: NCT02371824
Title: Study of Normal Hip and Lumbar Bone Marrow With Dynamic Contrast Enhancement Magnetic Resonance Imaging
Acronym: PERFOS
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_47; 2013-A01708-37 (Other: ID-RDB number, ANSM)
Record Dates: First submitted 2015-01-05; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Bone Marrow
Keywords: Magnetic Resonance Imaging; Bone Marrow; Hip; Lumbar Vertebrae

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MRI Sequence
  Interventions: Other: MRI sequence

INTERVENTIONS:
Other: MRI sequence — One supplementary MRI sequence Dynamic Contrast Enhancement (DCE) was added to the clinical protocol.
  Other Names: Supplementary MRI sequence

SUMMARY:
DCE-MRI were performed in sixty adults (hips and lumbar spine). For each region of interest studied, the investigators determined the morphology of each time-concentration curve (TCC) and calculated semi-quantitative and pharmacokinetic parameters: initial slope (IS), area under the curve (AUC), time to peak (TTP), Ktrans, Kep and Ve. Clinical data were collected anamnestically.

DETAILED DESCRIPTION:
MRI protocol Patients were examined on a 3T MR scan (Ingenia, Philips Healthcare, The Netherlands). Conventional sequences were acquired depending on the clinical problem. A T1 spin echo sequence imaged the right hip in the coronal plane. A previously described Dynamic 3D T1 Spoiled Gradient Echo covered the right hip (8). Its main features were as follows. 94 axial slices covered a Field of View (FOV) of 228 x 130 x 169 mm. TR, TE, flip angle and bandwidth per pixel were respectively 4.5 and 2.1 ms, 10°, 389 Hz. Acquisition and reconstruction matrix were 64 x 66 and 128 x 128 respectively. Temporal resolution was 13.5 seconds.

Three variable flip angles (VFA) sequences (3°, 10° and 17°) were acquired before injection. Each acquisition lasted 55 seconds. Five baseline scans were acquired. 0.1 mmol/kg of gadoteric acid (DOTAREM, Guerbet, France) were injected at the beginning of the sixth scan at a rate of 2.5ml/sec followed by 20cc of saline flush. Twenty dynamic scans were collected. Total examination time was 9 minutes.

Post-processing The investigators analyzed DCE images with the open-source software Osirix and DCE tool software (http://kyungs.bol.ucla.edu/software/DCE_tool/DCE_tool.html). A ROI was deposed in the common femoral artery to determine Arterial Input Function. T1 map was calculated from VFA acquisitions. The precise r1 relaxivity (3.4) of the contrast agent was introduced. These elements were used to calculate the time / gadolinium concentration curve. Tofts model was used.

The morphology of the curve was assessed visually according to the description made by van Rijswik (10). For each ROI, semi-quantitative and pharmacokinetic parameters were calculated: initial slope (IS), area under the curve (AUC), time to peak (TTP), transfer constant (Ktrans), rate constant (Kep) and extravascular-extracellular space volume (Ve). IS calculation included points 5 to 15. AUC and TTP were calculated from points 5 to 25. Parametric maps were obtained for the illustration of this work, but were not used for the analysis itself in order to avoid bias in the deposition of ROIs.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* patients who requires MRI examination of the hip or sacro-iliac joints
* patients who required a gadolinium injection for the clinical needs were included.
* normal appearing bones on MR images.

Exclusion Criteria:

* Patients under 18 years old,
* pregnant women, prisoners,
* patients unable to give informed consent,
* patients very painful and non-cooperative patients,
* Absolute contraindication to 3Tesla MRI (pacemaker, implantable pacemaker, metallic foreign body intraorbital)
* patients with previous or current history of hip, neoplastic, inflammatory or hematologic diseases, known osteoporosis or osteopenia, hip orthopedic hardware, chronic renal failure, known hyperparathyroidism, known acute or chronic inflammatory syndrome.
* abnormalities of the hip bones were seen on MR images, the patient was not included.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients referred to the musculoskeletal imaging department for a MRI examination of the hip or sacro-iliac joints with normal appearing bones on MR images.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Measure of transfer constant (Ktrans) | On the day of the visit
  This measure reflecting tissular perfusion is made in all the regions of interest.
Measure of rate constant (Kep) | On the day of the visit
  This measure reflecting tissular perfusion is made in all the regions of interest.
Measure of extra-vascular extra-cellular space (Ve) | On the day of the visit
  This measure reflecting tissular perfusion is made in all the regions of interest.
Measure of the initial slope (IS) of the Time-Concentration Curves | On the day of the visit
  This measure reflecting tissular perfusion is made in all the regions of interest.
Measure of the area under the curve (AUC) on the Time-Concentration Curves | On the day of the visit
  This measure reflecting tissular perfusion is made in all the regions of interest.
Measure of the time to peak (TTP) on the Time-Concentration Curves | On the day of the visit
  This measure reflecting tissular perfusion is made in all the regions of interest.

SECONDARY OUTCOMES:
Gender ratio | On the day of the visit
  In all the regions of interest, we sought for statistical correlation with the perfusion parameters listed as primary outcome measurements.
Age ratio | On the day of the visit
  In all the regions of interest, we sought for statistical correlation with the perfusion parameters listed as primary outcome measurements.
body mass index | On the day of the visit
  In all the regions of interest, we sought for statistical correlation with the perfusion parameters listed as primary outcome measurements.
number of smokers | On the day of the visit
  In all the regions of interest, we sought for statistical correlation with the perfusion parameters listed as primary outcome measurements.
number of alcohol consumers | On the day of the visit
  In all the regions of interest, we sought for statistical correlation with the perfusion parameters listed as primary outcome measurements.
number of participants with diabetes | On the day of the visit
  In all the regions of interest, we sought for statistical correlation with the perfusion parameters listed as primary outcome measurements.
number of participants with hypertension | On the day of the visit
  In all the regions of interest, we sought for statistical correlation with the perfusion parameters listed as primary outcome measurements.
number of participants with hypercholesterolemia | On the day of the visit
  In all the regions of interest, we sought for statistical correlation with the perfusion parameters listed as primary outcome measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Anne COTTEN, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hospital Center Roger Salengro, Lille, France